CLINICAL TRIAL: NCT02306785
Title: An Open Label, Single-site Pharmaco-Scintigraphic Study in Healthy Subjects and Patients With Active Ulcerative Colitis With Radio-labelled TP05-tablets to Evaluate the Gastrointestinal Transit and Release Profiles of Two Different Formulations (and Amendment)
Brief Title: TP0502-Pharmaco-Scintigraphic-Study and Amendment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TP0502 + A
Record Dates: First submitted 2014-10-15; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formulation D (Experimental): TP05 Coating D
  Interventions: Drug: TP05 Coating D
- Formulation E (Experimental): TP05 Coating E
  Interventions: Drug: TP05 Coating E
- Formulation H (Experimental): TP05 Coating H
  Interventions: Drug: TP05 Coating H

INTERVENTIONS:
Drug: TP05 Coating D — One radio-labelled tablet given to subjects
  Other Names: Mesalazine
  Arms: Formulation D
Drug: TP05 Coating E — One radio-labelled tablet given to subjects
  Other Names: Mesalazine
  Arms: Formulation E
Drug: TP05 Coating H — One radio-labelled tablet given to subjects
  Other Names: Mesalazine
  Arms: Formulation H

SUMMARY:
This is a Phase I, open-label, single-site trial to evaluate the drug release, using scintigraphic images and mesalazine plasma levels (PK) in healthy subjects and patients with mildly active UC. Overall, nine [9] subjects per prototype coating (a total of 18) will be evaluated. Four [4] healthy subjects and five [5] patients will be administered one [1] radio-labelled tablet of either formulation D or formulation E, respectively.

Amendment: Overall, nine [9] subjects/patients will be evaluated. Four [4] healthy subjects and five [5] patients will be administered one [1] radio-labelled tablet of this new third improved formulation H.

In order to keep the number of patients low, recruitment of patients will be stopped when obtaining at least 3 patients with evaluable scintigraphic images. Healthy volunteers will then be recruited to achieve a full set of participants (n=9 per Arm).

ELIGIBILITY:
Inclusion Criteria:

Main criteria for inclusion of healthy subjects include:

1. Healthy subjects, male or non-pregnant, non-lactating females, between 18 and 55 years old. Females of child bearing potential must have a negative serum pregnancy test prior to the intake of study drug, and must use a hormonal (oral, implantable or injectable) or a double barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
2. Ability of subject to participate fully in all aspects of this clinical trial.
3. Written informed consent must be obtained and documented.

Main criteria for inclusion of patients with mildly active Ulcerative Colitis (UC):

1. Male or non-pregnant, non-lactating females, between 18 and 55 years old. Females of child bearing potential must have a negative serum pregnancy test prior to the intake of study drug, and must use a hormonal (oral, implantable or injectable) or a double barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
2. UC patients with occasional streaks of blood in the stool during the past week
3. UC patients with a stool frequency of 1-2/day > normal
4. UC patients whose activity of disease is considered mild by his/her treating gastroenterologist
5. Ability of patient to participate fully in all aspects of this clinical trial
6. Written informed consent must be obtained and documented

Exclusion Criteria:

Main criteria for exclusion of healthy subjects include:

1. Participating in a clinical study involving investigational drugs or dosage forms within the previous 30 days.
2. History of alcohol or drug abuse.
3. Radiation exposure from clinical trials, including that from the present study and from diagnostic X-ray but excluding background radiation, exceeds 5 mSv (milli-Sievert) in the last five years. No subject whose occupational exposure is monitored will participate in the study.
4. Any nuclear medicine procedure prior to study day 1 that might interfere with the scintigraphic images that are acquired.
5. Clinically significant abnormal biochemistry, haematology or urinalysis:

   * White blood count <3 x 109/L and >8 x 109/L
   * Lymphocyte count < 0.85 x 109/L
   * Haemoglobin < 110g/L
   * Platelet count < 125 x 109/L or > 600 x 109/L
   * Alanine-Aminotransferase (ALT) or Aspartate-Aminotransferase (AST) > 2x upper limit of normal
   * Alkaline Phosphatase > 2x upper limit of normal
   * Serum Creatinine > upper limit of normal
6. History of gastrointestinal surgery, with the exception of appendectomy unless it was performed within the previous 12 months.
7. History of cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome (within the previous 12 months).
8. Acute diarrhoea or constipation in the 14 days before the predicted first study day. If screening occurs >14 days before first study day, this criterion is to be determined on the first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day.
9. History of adverse reaction or allergy to aspirin, mesalazine or other salicylates.
10. Donation of blood within the previous three months.
11. Positive HBV-Antigen (Hepatitis-B), HCV-Antibody (Hepatitis-C) or HIV-antibody (Human Immunodeficiency Virus) result.
12. Over-the-counter (OTC) and prescription medication (including laxatives, vitamins and natural herbal remedies) between screening visit (visit 1) and completion of the study. Occasional paracetamol or acetyl-salicylic acid is permitted.
13. Failure to satisfy the Principal Investigator to participate for any other reason.

Main criteria for exclusion of UC patients include:

The patients will only be included in the study if they do not meet any of the following criteria:

1. Participating in a clinical study involving investigational drugs or dosage forms within the previous 30 days.
2. History of alcohol or drug abuse.
3. Radiation exposure from clinical trials, including that from the present study and from diagnostic X-ray but excluding background radiation, exceeds 5mSv in the last twelve months. No patient whose occupational exposure is monitored will participate in the study.
4. Any nuclear medicine procedure prior to study day 1 that might interfere with the scintigraphic images that are acquired.
5. Clinically significant abnormal biochemistry, haematology or urinalysis:

   * White blood count <3 x 109/L and >8 x 109/L
   * Lymphocyte count < 0.85 x 109/L
   * Haemoglobin < 110g/L
   * Platelet count < 125 x 109/L or > 600 x 109/L
   * ALT, AST, total Bilirubin or alkaline phosphatase > 2 times the upper limit of normal
   * Serum Creatinine > 1.5 times the upper limit of normal
6. History of gastrointestinal surgery, with the exception of appendectomy unless it was performed within the previous 12 months.
7. History of cardiovascular, renal, hepatic, respiratory, peptic ulceration, gastrointestinal bleedings, Crohn's disease or Irritable Bowel Syndrome (within the previous 12 months) or any other disease which in the opinion of the investigator may interfere with the patient's ability to comply with the study procedures
8. Severe UC defined by the following criteria:

   ≥ 6 bloody stools daily with one or more of the following
   * oral temperature > 37.8°C
   * pulse > 90/min
   * hemoglobin < 100 g/L
9. History of adverse reaction or allergy to aspirin, mesalazine or other salicylates.
10. Donation of blood within the previous three months.
11. Positive HBV-Antigen, HCV-Antibody or HIV-antibody result.
12. Unwilling to stop oral or rectal mesalazine treatment on the treatment day if on mesalazine treatment before enrolment
13. History of colectomy or partial colectomy
14. History of dysplasia in colonic biopsies
15. Failure to satisfy the Principal Investigator to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Tablet release | 3 days

SECONDARY OUTCOMES:
Maximal Plasma concentration (Cmax) | 3 days
Time to reach Cmax (Tmax) | 3 days
Area under the concentration time-curve | 3 days
Elimination rate konstant (k) | 3 days
Lag time (T-lag) | 3 days